CLINICAL TRIAL: NCT02426658
Title: A Pilot Study Evaluating Pemetrexed in ECOG Performance Status 3 Patients With Stage IV Non-squamous Non-small Cell Lung Cancer
Brief Title: Pemetrexed Disodium in Treating Patients With Stage IV Non-small Cell Lung Cancer and ECOG Performance Status 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00032417; NCI-2015-00596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 62115; CCCWFU # 62115 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-08

CONDITIONS: Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pemetrexed disodium) (Experimental): Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Quality-of-Life Assessment and Laboratory Biomarker Analysis.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Other: Quality-of-Life Assessment — QOL studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot phase II trial studies how well pemetrexed disodium works in treating patients with stage IV non-small cell lung cancer and an Eastern Cooperative Oncology Group (ECOG) performance status of 3. Performance status means how well patients are able to perform daily activities and care for themselves. Patients with a performance status of 3 have a limited ability to move around. Currently, only patients who are able to perform most of their daily activities may receive chemotherapy, due to the side effects it may cause. Pemetrexed disodium causes fewer side effects than many chemotherapy drugs and may help treat patients with stage IV non-small cell lung cancer and a lower performance status.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of single agent pemetrexed (pemetrexed disodium) on tumor progression in ECOG performance status 3 patients with stage IV non-squamous histology non-small cell lung cancer in a single arm pilot study.

II. To evaluate the effect of single agent pemetrexed on quality of life in ECOG performance status 3 patients with stage IV non-squamous histology non-small cell lung cancer in a single arm pilot study.

SECONDARY OBJECTIVES:

I. To evaluate toxicity associated with single agent pemetrexed on tumor progression in ECOG performance status 3 patients with stage IV non-squamous histology non-small cell lung cancer in a single arm pilot study.

OUTLINE:

Patients receive pemetrexed disodium intravenously (IV) over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days and then every 6 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed Stage IV non-squamous histology non-small cell lung cancer
* ECOG performance status of 3
* Sensitizing epidermal growth factor receptor (EGFR), anaplastic lymphoma receptor tyrosine kinase (ALK) and ROS proto-oncogene 1, receptor tyrosine kinase (ROS-1) mutations are either negative or unknown
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Creatinine clearance >= 45 mL/min
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document
* Ability to understand and complete the European Organization for Research and Treatment of Cancer (EORTC) quality of life (QOL) instruments

Exclusion Criteria:

* Patients who have previously received chemotherapy for non-small cell lung cancer, or have received radiotherapy within 2 weeks prior to entering the study, or who have not recovered from adverse events due to treatment more than 2 weeks earlier
* Patients whose tumors are positive for the sensitizing EGFR mutation
* Patients whose tumors are positive for the sensitizing ALK fusion
* Patients whose tumors are positive for the sensitizing ROS-1 fusion
* Patients may not be receiving any other investigational agents
* Patients with symptomatic or recurrent brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pemetrexed
* Pregnant women are excluded from this study; breastfeeding should be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grant, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pemetrexed Disodium)
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Patient expired before treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pemetrexed Disodium)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life (QOL), Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (QLQ-C30) and QLQ-Lung Cancer 13-item (LC13)
Description: Quality of life will be assessed at each treatment time (i.e. every three weeks). A longitudinal mixed models analysis will be used to look at QOL over the time course. A paired t-test will also be calculated to see if the average change is more than 0 (worsening) versus a two-sided alternative that the difference is 0 or better. Score range from 0-100 (1 = not at all, 2 = a little, 3 = quite a bit, or 4 = very much). The higher the score, the greater the change in the quality of life for the worse.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment (Pemetrexed Disodium)
Number analyzed (Participants) | 13
score on a scale
  Baseline | 51.2821 (6.6951)
  12 weeks | 58.3333 (17.0693)
Statistical Analysis 1: Comparison: Treatment (Pemetrexed Disodium); Test type: Superiority; p = 0.7044, Mixed Models Analysis

2. Primary Outcome: Time to Tumor Progression
Description: It will be determined whether each patient has a progression (or dies) before or after 12 weeks. A 95% exact (Clopper Pearson) confidence interval will then be around the proportion with PFS greater than or equal to 12 weeks. If this confidence interval includes 50% then that would provide evidence that the therapy is potentially promising. If the upper bound of the confidence interval does not include 50% then this would indicate that the treatment may not be promising for patients. In addition, a Kaplan Meier survival curve will be constructed to describe the time to progression data.
Time Frame: The duration of time from the start of treatment to the time of progression, death, or date of last contact, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pemetrexed Disodium)
Number analyzed (Participants) | 12
months | 2.0 [1.0 to 10.7]

3. Secondary Outcome: Incidence of Hematologic Toxicity, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The number and type of toxicities observed during this protocol will be estimated, focusing on unexpected grade 3 or higher toxicities. No formal statistical tests will be done on these estimates.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pemetrexed Disodium)
Number analyzed (Participants) | 13
Participants
  Anemia | 13
  CD4 lymphocyte decreased | 3
  Febrile neutropenia | 1
  Leukocytosis | 1
  Lymphocyte count decreased | 9
  Neutrophil count decreased | 11
  Platelet count decreased | 10
  White blood cell count decreased | 10

4. Secondary Outcome: Overall Survival
Description: Examined by estimating a Kaplan-Meier survival curve using all patients enrolled.
Time Frame: The duration of time from the start of treatment to date of death or date of last contact, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pemetrexed Disodium)
Number analyzed (Participants) | 13
months | 2.4 [1.0 to 10.7]

5. Secondary Outcome: Response Rate
Description: Response rate will be estimated every 6 weeks for patients, and these estimates will be presented with confidence intervals.
Time Frame: Up to 2 years
Population: Four patients died prior to the 2nd cycle of treatment when this measure was evaulated.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pemetrexed Disodium)
Number analyzed (Participants) | 9
Participants
  Partial response | 1
  Stable disease | 6
  Progressive disease | 2

ADVERSE EVENTS:
Time Frame: 30 days after the last study is administered
Arm/Group | Treatment (Pemetrexed Disodium)
All-Cause Mortality (participants affected / at risk) | 4/13
Serious Adverse Events (participants affected / at risk) | 12/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pemetrexed Disodium) (N=13)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Death, NOS (General disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pemetrexed Disodium) (N=13)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 10 (18)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
CD4 lymphocytes decreased (Investigations) | 3 (4)
Cardiac disorders, other (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Creatinine increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Edema limbs (General disorders) | 3 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
General disorders and administration site disorders, other (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (6)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (26)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 9 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Investigations, other (Investigations) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Lymphocyte count decreased (Investigations) | 7 (11)
Metabolism and nutrition disorders, other (Metabolism and nutrition disorders) | 1 (1)
Mucositis, oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (7)
Neutrophil count decreased (Investigations) | 6 (6)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Platelet count decreased (Investigations) | 7 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02426658/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT02426658/ICF_001.pdf